CLINICAL TRIAL: NCT05745935
Title: Role of Local Skin Incision Infiltration by Oxytocin On Wound Healing of Caesarean Section Scar in Primiparous Women A Double Blind Randomized Controlled Study
Brief Title: Role of Local Skin Incision Infiltration by Oxytocin On Wound Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Assem Anour
Record Dates: First submitted 2023-02-12; First posted 2023-02-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Wound Heal; Scar; Previous Cesarean Section
Keywords: wound healing; Oxytocin; caesarean Section scar; wound complications
MeSH Terms: conditions — Cicatrix | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): About 50 Patients Will receive 20 units of local oxytocin infiltration before skin closure . 10 units of oxytocin will be infiltrated at the upper skin edge and 10 units of oxytocin will be infilterated at the lower skin edges at equal intervals of 2 cm in between infiltration points.
  Interventions: Drug: Oxytocin
- Group B (Experimental): About 50 Patients Will receive the 10 units of local oxytocin infiltration before skin closure . 5 units will be infiltrated at the upper skin edge and 5 units will be infiltrated at the lower skin edge at equal intervals of approximately 2 cm in between infiltration points.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — This study will include 100 elective cesarean section in parous women who will be randomized into two groups each of 50 patients,
  Other Names: Syntoinon

SUMMARY:
caesarean section rate in Egypt has reached about 60% between primgravidae.

Wound complications are of the most common morbidities following cesarean section. The prevalence of wound infection and disruption after cesarean has been reported as 3-15%, averagely speaking 6% and 2-42% in various studies.

These complications affect mother's quality of life due to stress, anxiety, delay in mother's ability and health recovery

DETAILED DESCRIPTION:
Nowadays, cesarean is one of the most common surgical interventions and its prevalence has increased in most countries in the recent years.

At present, all efforts are focused on the early and effective healing of caesarean skin wound and its associated complications.

There is a wide range of topical and systemic treatments for the management of caesarean skin incision. Topical treatments have side effects and hence are not considered as the treatment of choice for such incisions.

Oxytocin is a Nonapeptide hormone of a cyclic six amino-acid structure and a tail of three amino acids, responsible for initiation of the milk ejection reflex and stimulating the uterine contractions.

However, other important roles of oxytocin include improvement of social life, exerting pain-relieving, anti anti-stress/anti-inflammatory and restorative effects, friendship and making social relationship with individual or group.

However, other important roles of oxytocin include improvement of social life, exerting pain-relieving, anti anti-stress/anti-inflammatory and restorative effects, friendship and making social relationship with individual or group.

In conclusion, oxytocin is linked to many different, sometimes opposite effects The intact cyclic molecule may act to initiate social interaction and associated psychophysiological effects, whereas linear oxytocin and C-terminal fragments may induce relaxation and anti-stress effects following social interaction.

In this way, the principal hormone oxytocin and its fragments may take part in a behavioral sequence, ranging from approach and interaction to calm and relaxation.

Linear fragments, with an exposed cysteine-residue, may exert anti-inflammatory and antioxidant effects and thereby contribute to the health-promoting effects of oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Primigravidae women,
* Age group from 20- 35 years old.
* Gestational age 37-41 weeks, and
* Elective caesarean section due to obstetrics indication.
* The patient signed an Informed Consent Form authorizing their inclusion

Exclusion Criteria:

* Multiparous women,
* Assisted vaginal delivery,
* Normal vaginal delivery,
* Emergency caesarean section,
* Preterm pre labour rupture of membrane,
* Primiparous women with age above 35 years old,
* Primiparous women with known connective tissue disease and
* Women suffering from chronic diseases such as diabetes, hypertension, cardiovascular diseases, psychiatric diseases, cancer
* Smoking Women

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Wound healing after Oxytocin injecton | from baseline to 6 days after the Cesarean operation
  Injection of the Oxytocin hormon in the cesarean wound before closing it during cesarean delivery and close watching for healing process.
Pain Relief | From base line to 6 hours postoperatively
  The effect of oxytocin on pain relief using pain score scale, numerical pain score scale from 0-10 where 0 is no pain, from 1-3 is mild pain,4-6 moderate pain and from 7-10 is severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Assem Anour, Professor, Principal Investigator — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al Amerya hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided